CLINICAL TRIAL: NCT05636683
Title: Evaluation of Bone Remodeling Markers Following Non-surgical Periodontal Therapy in Periodontitis Patients (Prospective Clinical Trial)
Brief Title: Bone Remodeling and Non-surgical Periodontal Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Firas Bashir Hashim Al-Taweel, Assistant Professor, University of Baghdad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 665622
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Periodontitis treated with Root surface debridement (Experimental): Immediately after inclusion in the study, the patient's examination with saliva sampling will be conducted as follows: At a base line visit (Zero time visit), subjects will be examined for clinical periodontal parameters, their saliva samples will be collected, and then receiving full scaling using ultrasonic device, and oral hygiene instructions and motivation. After one week, the same clinical parameters, saliva sampling will be taken, and received full root surface debridement (RSD) using curette hand instruments (Gracey, USA) (First visit). One month and three months after first visit, the same clinical measurements, saliva will characterize as second and third visits, respectively.
  Interventions: Procedure: Root surface debridement

INTERVENTIONS:
Procedure: Root surface debridement — subjects will be examined for clinical periodontal parameters, their saliva samples will be collected, and then receiving full scaling using ultrasonic device, and oral hygiene instructions and motivation. After one week, the same clinical parameters, saliva sampling will be taken, and received full root surface debridement (RSD) using curette hand instruments (Gracey, USA) (First visit). One month and three months after first visit, the same clinical measurements, saliva will characterize as second and third visits, respectively.

SUMMARY:
Previous studied have investigated the pathophysiological role and expression of Cathepsin K (Ctsk) , receptor activator of the NF-κB ligand (RANKL) and periostin in active periodontitis and peri-implantitis lesions. However, the potential influence of non-surgical periodontal therapy including scaling and root planning on the bone remodeling markers level over different trial times have not well determined. Thus, the current research is conducted to address this influence. Thus, the research question will be: In patients with periodontitis, does the level of bone remodeling markers altered after successful NSPT during different healing time periods?

ELIGIBILITY:
Inclusion Criteria:

1. Both males and females.
2. Unstable periodontitis.
3. No previous periodontal treatment is conducted during the past 6 months.
4. Good general health without history of any systemic diseases.
5. Present with at least 20 teeth.
6. Non-smokers.

Exclusion Criteria:

1. Subjects have any intraoral plaque retentive factors such as those wearing partial denture, crown and bridges, and orthodontic appliances.
2. Subjects receiving antibiotic therapy during the previous 3 months.
3. Pregnant or lactating women.
4. Smokers.
5. Not willing to participate or continue to conduct the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Bone remodeling markers including salivary RANKL | At a base line visit (Zero time visit), After one week (first visit), and One month and three months after first visit
  To investigate the alterations in the level of salivary RANKL pg/ml following Non-surgical periodontal therapy in unstable periodontitis patients during different healing time periods.
Bone remodeling markers including salivary Cathepsin k | At a base line visit (Zero time visit), After one week (first visit), and One month and three months after first visit
  To investigate the alterations in the level of salivary Cathepsin k pg/ml following Non-surgical periodontal therapy in unstable periodontitis patients during different healing time periods.
Bone remodeling markers including salivary periostin | At a base line visit (Zero time visit), After one week (first visit), and One month and three months after first visit
  To investigate the alterations in the level of salivary periostin pg/ml following Non-surgical periodontal therapy in unstable periodontitis patients during different healing time periods.

SECONDARY OUTCOMES:
Clinical periodontal parameters including Bleeding on probing | At a base line visit (Zero time visit), After one week (first visit), and One month and three months after first visit
  To measure Clinical periodontal parameters including Bleeding on probing following Non-surgical periodontal therapy in unstable periodontitis patients during different healing time periods.
Clinical periodontal parameters including probing pocket depth | At a base line visit (Zero time visit), After one week (first visit), and One month and three months after first visit
  To measure Clinical periodontal parameters including probing pocket depth following Non-surgical periodontal therapy in unstable periodontitis patients during different healing time periods.
Clinical periodontal parameters including clinical attachment loss | At a base line visit (Zero time visit), After one week (first visit), and One month and three months after first visit
  To measure Clinical periodontal parameters including clinical attachment loss following Non-surgical periodontal therapy in unstable periodontitis patients during different healing time periods.

CONTACTS AND LOCATIONS:
Overall Officials: Firas B. Al-Taweel, PhD, Study Director — Periodontics department, College of Dentistry/University of Baghdad
Locations (1):
- College of Dentistry, University of Baghdad, Baghdad, Iraq